CLINICAL TRIAL: NCT04578730
Title: A Prospective, Observational (Non-interventional), International Study to Assess Conservative Treatments Effectiveness in Acute Phase of Hemorrhoidal Disease
Brief Title: aCute HemORrhoidal Disease evALuation International Study
Acronym: CHORALIS
Status: Completed | Type: Observational
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Other Study IDs: DIM-05682-006-INT
Record Dates: First submitted 2020-09-15; First posted 2020-10-08 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Hemorrhoids
Keywords: observationnal; QoL
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to assess in real-life setting the effectiveness of conservative treatments on signs, symptoms and quality of life in patients consulting for hemorrhoids in acute phase of the disease

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Patient consulting for symptomatic acute phase of hemorrhoidal disease
* Confirmed diagnosis of hemorrhoidal disease

Exclusion Criteria:

* Patient consulting for emergency not related to hemorrhoidal disease;
* Patient currently taking any treatment for hemorrhoidal disease;
* Any anorectal procedure or surgery planned during the study ;
* Anorectal procedure or surgery performed or incomplete convalescence following anorectal procedure/surgery;
* Known present perianal sepsis, inflammatory bowel disease, colorectal malignancy, pre-existing sphincter injury, diseases of the anal canal;
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from hemorrhoidal disease in the acute phase
Sampling Method: Non-Probability Sample
Enrollment: 3592 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Global improvement | Week 4
  Measured by Patient Global Impression of Change (PGIC) scale, and time to improvement.
Signs and symptoms severity: pain, discomfort, bleeding, prolapse, swelling, itching, and soiling | Week 4
  Measured by VAS (Visual analogue scale) and questioning with 4 points rate
Quality of Life | Week 4
  Measured by HEMO-FISS QoL

CONTACTS AND LOCATIONS:
Locations (1):
- Servier Affaires Medicales, Suresnes, France